CLINICAL TRIAL: NCT04301050
Title: Learning Yoga to eNhance Cancer Survivorship
Acronym: LYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Elizabeth Addington, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00209987
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Cancer
Keywords: Young Adult; Cancer Survivor
MeSH Terms: conditions — Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Intervention (Experimental): Participants will complete 8-week course (75-minute, weekly yoga classes) delivered online via videoconferencing software. Participants will complete patient-reported outcomes at baseline (prior to class 1) and post-intervention (after class 8), as well as post-intervention measures of feasibility/acceptability.
  Interventions: Other: Yoga Intervention

INTERVENTIONS:
Other: Yoga Intervention — Weekly 75-minute yoga classes.
  Other Names: Yoga

SUMMARY:
This study aims to conduct a single-arm pilot test of online yoga classes for young adult cancer survivors (YACS). Study hypotheses are that LYNC will be feasible (enrollment of > 50% of eligible) and acceptable (75% attendance at all sessions). In addition, analyses of preliminary efficacy outcomes will examine whether participants report potential improvements in psychosocial and physical wellbeing.

DETAILED DESCRIPTION:
This study will recruit YACS (n=30) for an 8-week course (75-minute yoga classes delivered once per week) delivered online via videoconferencing software such as Zoom or Bluejeans. During yoga classes, all participants will be able to see one another, to simulate the group experience of being in an in-person class. Participants will complete patient-reported outcomes of physical and psychosocial wellbeing at baseline (prior to class 1) and post-intervention (after class 8), as well as post-intervention measures of feasibility/acceptability (e.g., ease of accessing online classes, satisfaction with yoga classes, helpfulness of online yoga, barriers/dislikes associated with online yoga). All surveys will be administered via REDCap. In addition, the investigators will compute rates of retention (% of consenting subjects who complete post-intervention assessment) and adherence (# of yoga classes attended).

ELIGIBILITY:
Inclusion Criteria:

* Age 25-39
* History of cancer diagnosed at age >18
* >2 months post-treatment for cancer
* Eastern Cooperative Oncology Group (ECOG) performance status (0-2)
* Access to internet-connected device with camera and capacity for full-screen display (e.g., laptop or desktop computer; tablet or smart phone with Air Play to full-size monitor)

Exclusion Criteria:

* Regular use of yoga (i.e., once or more per week) since cancer diagnosis/treatment
* Unable to complete forms and yoga classes in English
* Adults who are cognitively impaired, pregnant, imprisoned or otherwise detained

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility | 9 months
  Enrollment rate of > 50% of eligible screened participants
Acceptability | 8 weeks
  Attendance rate: >75% of classes, on average

SECONDARY OUTCOMES:
Change in Health Behaviors | [Baseline, 8 week]
  Health behaviors are measured with a 10-item scale adapted from investigators' prior research. Items allow for calculation of body mass index (based on self-reported height and weight), determination of the amount of physical activity per week, and indicators of diet quality. Items are based on American Cancer Society and National Comprehensive Cancer Network guidelines for health behaviors in cancer survivors.
Change in Interoceptive Awareness | [Baseline, 8 week]
  As measured by a change in the body listening and trusting sub scales of the Multidimensional Assessment of Interoceptive Awareness (Version 2). Scores on this scale range from 0-5, with higher scores indicating greater interoceptive awareness.
Change in Depression | [Baseline, 8 week]
  As measured by PROMIS SF (Patient Reported Outcomes Measurement Information System Short Form) v1.0 - Depression 4a
Change in Anxiety | [Baseline, 8 week]
  As measured by PROMIS SF v1.0 - Anxiety 4a
Change in Sleep Disturbance | [Baseline, 8 week]
  As measured by PROMIS SF v1.0 - Sleep Disturbance 4a
Change in Fatigue | [Baseline, 8 week]
  As measured by PROMIS SF v1.0 - Fatigue 7a
Change in Pain Intensity | [Baseline, 9 week]
  As measured by PROMIS Scale v1.0 - Pain Intensity 3a PROMIS SF v1.0 - Fatigue 7a
Change in Pain Interference | [Baseline, 8 week]
  As measured by PROMIS SF v1.0 - Pain Interference 6b
Change in Physical Function | [Baseline, 8 week]
  As measured by PROMIS SF v2.0 - Physical Function 4a PROMIS SF v2.0 - Physical Function 4a
Change in Positive Affect | [Baseline, 8 week]
  As measured by PROMIS SF v1.0 - Positive Affect 15a PROMIS SF v1.0 - Positive Affect 15a
Change in Social Isolation | [Baseline, 8 week]
  As measured by PROMIS SF v2.0 - Social Isolation 8a

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Addington, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No